CLINICAL TRIAL: NCT00257985
Title: Glyceryl-Trinitrate-Induced Headache in Patients With Familial Hemiplegic Migraine Type 1 and 2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Danish Headache Center (Other)
Collaborators: EUROHEAD (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Educational/Counseling/Training
Other Study IDs: FHM-GTN 2005
Record Dates: First submitted 2005-11-22; First posted 2005-11-24 (Estimated); Last update posted 2006-08-01 (Estimated); Status verified 2005-11

CONDITIONS: Familial Hemiplegic Migraine Type 1 and 2; Healthy Volunteers
Keywords: Familial hemiplegic migraine type 1 and 2; GTN; middle cerebral artery; superficial temporal artery; headache; genotype
MeSH Terms: conditions — Hemiplegic migraine, familial type 1; Headache

INTERVENTIONS:
Drug: GTN

SUMMARY:
The aim of the present study is to explore functional consequences of migraine gene mutations on their responses to GTN infusion.

DETAILED DESCRIPTION:
Glyceryl trinitrate (GTN) induces migraine attacks indistinguishable from spontaneous attacks in approximately 80% of migraine sufferers. After systemic administration GTN is transformed to nitric oxide (NO). Treatment of spontaneous migraine attacks with an inhibitor of NO is effective in 60% of patients. These data show that NO is involved in both initiation and maintenance of migraine attack.

The consequence of migraine gene mutations on relevant migraine pathways has never been tested. The aim of the present study is to explore functional consequences of migraine gene mutations on their responses to GTN infusion. The project will improve our understanding of the neurobiology of migraine and stimulate development of new treatment targets.

ELIGIBILITY:
Inclusion Criteria:

Patients: Diagnosis of familial hemiplegic migraine (IHS-classification criteria) caused by mutations in the CACNA1A gene and the ATP1A2 gene.

Controls: healthy volunteers

Exclusion Criteria:

Controls: No primary headache in their own history

Patients and controls:

* A history of cerebrovascular disease and other CNS- disease
* A history of serious somatic and mental disease
* A history suggesting ischaemic heart disease
* A history of hypo- or hypertension
* Daily intake of medication apart from oral contraceptives
* Abuse of alcohol or medicine (opioid analgesics).
* Pregnant or breastfeeding women.

On the study day:

* No intake of a simple analgesic in the previous 48 hours
* No headache in the previous 48 hours

Min Age: 0 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30
Dates: Start 2005-04; Study Completion 2006-03

PRIMARY OUTCOMES:
headache and associated symptoms , blood flow velocity of the middle cerebral artery, diameter of the superficial temporal artery

SECONDARY OUTCOMES:
MAP, HR

CONTACTS AND LOCATIONS:
Overall Officials: Jakob Møller Hansen, MD, Principal Investigator — Danish Headache Center
Locations (1):
- Danish Headache Center, University of Copenhagen, Department of Neurology, Glostrup Hospital, Glostrup, Copenhagen, Denmark